CLINICAL TRIAL: NCT00691756
Title: A Comparison of Cold Blood Versus Cold Crystalloid Renal Perfusion for Prevention of Acute Renal Failure Following Thoracoabdominal Aortic Aneurysm Repair: A Randomized Study
Brief Title: A Comparison of Renal Perfusion in Thoracoabdominal Aortic Aneurysm (TAAA) Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Gillson-Longenbaugh Foundation (Other); Texas Heart Institute (Other)
Responsible Party: Principal Investigator, Scott Lemaire, Professor, Surgery/Cardio/Thoracic Surg., Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-9764
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Renal Failure
Keywords: renal failure; thoracoabdominal aortic aneurysm repair; cold crystalloid; cold blood; renal perfusion
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Cold blood renal perfusion
  Interventions: Procedure: Cold blood renal perfusion
- 2 (Active Comparator): Cold crystalloid renal perfusion
  Interventions: Procedure: Cold crystalloid renal perfusion

INTERVENTIONS:
Procedure: Cold blood renal perfusion — Both kidneys receive intermitent perfusion with cold (4 degrees C) autologous blood during thoracoabdominal aortic aneurysm repair.
  Arms: 1
Procedure: Cold crystalloid renal perfusion — Both kidneys receive intermittent perfusion with cold (4 degrees C) lactated Ringer's solution during thoracoabdominal aortic aneurysm repair. This is the standard renal perfusion technique in our practice.
  Arms: 2

SUMMARY:
The purpose of this randomized trial was to determine whether renal perfusion with cold blood provides better protection against renal ischemia than perfusion with cold crystalloid in patients undergoing TAAA repair with left heart bypass.

DETAILED DESCRIPTION:
Despite improvements in surgical techniques and postoperative care, renal dysfunction has consistently remained a significant and potentially lethal complication after thoracoabdominal aortic aneurysm (TAAA) repair. In an attempt to alleviate postoperative renal failure and its associated mortality, several techniques and intraoperative strategies have been used including: intraoperative administration of diuretics, steroids, or prostaglandins; minimization of ischemic times; renal hypothermia with cold crystallid solutions; selective warm (normothermic) blood perfusion as part of a left heart bypass (LHB) system; and hemodilution. However, despite the use of adjuvant techniques, the incidence of renal failure after TAAA repair still ranges from 3% to 27%. One of the techniques mentioned above involves cold crystalloid renal artery perfusion. This method aims to reduce metabolic needs of the renal system by inducing local hypothermia. Because oxygen consumption decreases 7% for each degree Celsius that temperature is reduced, the metabolic needs of tubular cells are reduced by almost 50% at 30 degrees Celsius. After the aorta is clamped and opened, the renal arteries are perfused with lactated Ringers solution (LR) that has been cooled to 4 degrees Celsius utilizing a roller pump to transport the LR through an appropriately cooled ice bath. This decreases the temperature of the kidneys to an average of 20 degrees Celsius. The volume of LR required to achieve this temperature ranges from 600 to 1800 ml. Renal cooling has been shown to preserve renal tissue as long as warm ischemic time is kept to a minimum. We recently compared renal artery cold crystalloid perfusion with normothermic blood perfusion in a randomized clinical trial involving 30 patients and discovered via multivariable analysis that cold LR was protective against acute postoperative renal dysfunction. In this study, we found that 62.5% of patients receiving normothermic blood perfusion developed acute postoperative renal dysfunction versus 21.4% in the cold LR group (p = 0.03). One method of renal protection not often used involves selective cold blood perfusion of the renal arteries. This technique also aims to reduce renal ischemic time during aortic cross-clamping and improve oxygenation to renal tissues; thereby, preventing reperfusion injury and organ dysfunction often associated with this operation. During aneurysm repair, left atrio-distal aortic bypass is performed using a centrifugal pump. Tubing connected to the distal end of this circuit passes through a container of ice allowing the perfusion of both renal arteries with cold blood. The flow rates into the renal arteries range from 100 to 450 ml/min. The celiac axis and superior mesenteric artery remain individually perfused in the standard fashion using normothermic blood. The best method of achieving renal protection remains unclear. Currently, normothermic blood and cold LR remain the two most commonly used methods of renal artery perfusion during TAAA repair. This randomized trial compared the effectiveness of two forms of renal artery perfusion, cold LR versus cold blood, to identify which method is more beneficial in the prevention of postoperative renal dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* age equal to or greater than 18
* planned extent II or III thoracoabdominal aortic aneurysm repair
* planned left heart bypass
* patient consent obtained

Exclusion Criteria:

* impaired left ventricular function
* impaired renal function
* prior thoracoabdominal aortic aneurysm repair
* pseudoaneurysm
* pre-existing liver disease
* free aortic aneurysm rupture
* inability to measure renal temperature
* extent I or IV thoracoabdominal aortic aneurysm repair

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2002-01; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Renal dysfunction | 10 postoperative days

SECONDARY OUTCOMES:
Renal injury (increase in urinary biomarkers) | 7 postoperative days

CONTACTS AND LOCATIONS:
Overall Officials: Scott A. LeMaire, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu D, Coselli JS, Johnson ML, LeMaire SA. Hepatopancreaticobiliary Values after Thoracoabdominal Aneurysm Repair. Aorta (Stamford). 2014 Aug 1;2(4):135-42. doi: 10.12945/j.aorta.2014.14-015. eCollection 2014 Aug. PMID 26798731
- [Result] Lemaire SA, Jones MM, Conklin LD, Carter SA, Criddell MD, Wang XL, Raskin SA, Coselli JS. Randomized comparison of cold blood and cold crystalloid renal perfusion for renal protection during thoracoabdominal aortic aneurysm repair. J Vasc Surg. 2009 Jan;49(1):11-9; discussion 19. doi: 10.1016/j.jvs.2008.08.048. Epub 2008 Nov 22. PMID 19028052